CLINICAL TRIAL: NCT00268021
Title: The Use of Automated Cardioverter Defibrillator in Children (AICD)
Brief Title: Automated Cardioverter Defibrillator in Children
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 04-082
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Disorders
Keywords: pediatric; biventricular pacemaker; automated implantable cardioverter defibrillator; AICD
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Automated implantable cardioverter defibrillators ,AICD, and Biventricular,BiV, Pacemakers have been shown in randomized trials to offer an advantage in adults with decreased ventricular ejection fraction, heart failure, spontaneous non-sustained ventricular tachycardia VT, inducible non-suppressible VT and the combination of low ejection fraction and prior myocardial infarction,14. Pediatric patients with a variety of different heart abnormalities are at high risk for life threatening arrhythmias and poor ventricular function or heart failure,16. Therefore, extrapolating this adult data, AICDs and BiV pacemakers have been used with increasing frequency in the pediatric and congenital heart disease population. Improvements in device size and lead design allows AICD and BiV implantation in the very young, in small size patients and in patients with complex cardiac anomalies,1. The use of BiV pacemakers and the patterns of AICD discharge are similar in young patients and in adults, suggesting that the risk of life threatening arrhythmia and heart failure are also similar,16. However, this patient population behaves differently from the adult population in the incidence of pacemaker complications, circadian arrhythmias,7, and more importantly, a relatively high incidence of complications related to AICD insertion, 8. There is a need for more studies to establish the risk-benefit ratio of these devices in the pediatric setting.

DETAILED DESCRIPTION:
This is a retrospective review of all the patients that had an AICD or BiV pacemakers inserted at Children's Healthcare of Atlanta at Egleston, Emory University, between January 1st, 1998 and July 30th, 2004. The goal of our study is to establish the prevalence of beneficial and adverse effects in the AICD and BiV patient population.

Demographic, clinical and electrophysiologic characteristics during the hospitalization as well as at follow-up will be obtained from the medical records and are summarized in the following tables Note: We defined infection as elevated temperature above 38.1 C associated with elevated WBC and positive cultures.

Appendix A

We plan to collect the following demographic information. Age Weight Delivery method Gestational age Weight at birth Delivery complications Cardiac anomalies Other anomalies

We plan to collect the following medical information/diagnoses. Indication Cardiac arrest Sustained ventricular tachycardia Inducible ventricular tachycardia Syncope Palpitations Severe hypertrophic cardiomyopathy Congenital heart disease Primary electrical disease Hypertrophic cardiomyopathy Idiopathic dilated cardiomyopathy

We will collect the following AICD information. Lead Transvenous Subcutaneous array Epicardial patches Generator type

We will collect the following outcomes information (AICD and BiV). Variable Appropriate discharge (AICD only) Inappropriate discharge (AICD only) Lead failure Overall survival Hospital Length of Stay Infection Blood transfusion/bleeding Hospital Re-admission Mortality/Morbidity information Cause of inappropriate AICD discharge/shock Long term complications

ELIGIBILITY:
Inclusion Criteria:

* patients with AICD inserted at Children's Healthcare of Atlanta
* patients with BiV pacemaker inserted at Children's Healthcare of Atlanta
* insertions between 1.1.1998 and 7.30.2004

Exclusion Criteria:

* those patients who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with AICD or BiV insertions
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: Kirk R Kanter, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States